CLINICAL TRIAL: NCT00884988
Title: The Efficacy of Lymphomyosot in the Treatment of Posttraumatic Edema Following Ankle Fracture, Pending Surgery: a Randomized, Double-blind, Placebo-controlled Study.
Brief Title: Lymphomyosot for Ankle Edema Following Fracture
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Study recruiter withdrew from study. Suspended until replacement found.
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Menachem Oberbaum, Director, Center for Integrative Complementary Medicine, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LYM.ANKLE.09
Record Dates: First submitted 2009-04-19; First posted 2009-04-21 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Ankle Injuries; Fracture
Keywords: ankle fracture; edema; surgical repair; homeopathy; lymphomyosot
MeSH Terms: conditions — Ankle Injuries; Fractures, Bone; Ankle Fractures; Edema | interventions — Lymphomyosot

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lymphomyosot (Active Comparator): homeopathic remedy
  Interventions: Drug: Lymphomyosot
- Placebo remedy (Placebo Comparator): identical in color, constituency and taste to true remedy
  Interventions: Drug: Placebo remedy

INTERVENTIONS:
Drug: Lymphomyosot — 20 drops X3/day, until discharge
  Arms: Lymphomyosot
Drug: Placebo remedy — 20 drops X3/day, until discharge
  Arms: Placebo remedy

SUMMARY:
Ankle fractures are invariably complicated by severe soft-tissue swelling which can significantly prevent surgical repair (open reduction and internal fixation - ORIF) of the fractured bone for up to two weeks. The delay in surgical treatment can increase the risk for local skin and bone complications, as well as for deep venous thrombosis. Lymphomyosot® is a non-prescription, homeopathic complex drug which has been used for more than 70 years throughout Europe and the U.S., primarily for tissue edema and swelling.

This is a randomized, placebo-controlled, double blind pilot study evaluating the effectiveness of homeopathic combination drug Lymphomyosot® compared to placebo treatment. The study will take place at the Shaare Zedek Medical Center in Jerusalem, Israel. Adult patients (age 18 years and older) admitted to the orthopedic department with acute ankle fractures which require ORIF repair will be assessed for inclusion in this study.

The primary outcome measure to be evaluated is the fracture-ORIF waiting period. Other measures to be evaluated are: peri-malleolar circumference; pain (as measured by NRS and analgesic use); duration of hospital stay; and complications such as poor wound healing, blisters, and the development of deep vein thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* patients with a fracture of the ankle requiring ORIF
* signed informed consent form.

Exclusion Criteria:

* refusal or inability to give informed consent
* bilateral fractures of the foot or ankle, open fractures, poly-trauma, contralateral limb amputation
* currently on anticoagulation therapy
* clinical indication for immediate surgery.
* ability to undergo surgery on the day of the fracture , or where soft-tissue edema was not the cause which prevented immediate surgery
* any additional injury that prevents partial weight-bearing.
* a concomitant fracture of another long bone in the ipsilateral leg
* if the patient suffers from a systemic disease such as diabetes, malignant tumor, severe peripheral vasculopathy, and/or metabolic disease
* concurrent participation in another study
* inability to comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-02; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
To compare the effect of Lymphomyosot on the duration of time from fracture to ORIF surgery, to placebo medication. | 3 weeks

SECONDARY OUTCOMES:
To compare the effect of Lymphomyosot® on the development of peri-malleolar edema following ankle fracture surgery, to placebo medication. | 3 weeks
To compare the effect of Lymphomyosot on pain following ankle fracture, to placebo medication. | 3 weeks
To compare the effect of Lymphomyosot on Hospitalization time between the verum and the placebo group. | 3 weeks
To compare the effect of Lymphomyosot on complication rate (wound healing disturbance, wound infection, blistering, deep vein thrombosis). | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Menachem Oberbaum, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel